CLINICAL TRIAL: NCT02328586
Title: Group Acupuncture for Pain
Acronym: GAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070-14
Record Dates: First submitted 2014-07-03; First posted 2014-12-31 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group Acupuncture (Experimental): Participants will then be invited to participate in an 8-week, group-based acupuncture treatment intervention delivered by a licensed acupuncturist. The group will meet weekly for 8 consecutive weeks, each session lasting about 75 minutes.
  Interventions: Other: Group Acupuncture

INTERVENTIONS:
Other: Group Acupuncture

SUMMARY:
This research project will test the feasibility and effectiveness of group acupuncture for the treatment of musculoskeletal pain (back pain, shoulder pain, neck pain and/or osteoarthritis).

DETAILED DESCRIPTION:
This research project will test the feasibility and effectiveness of group acupuncture for the treatment of musculoskeletal pain (back pain, shoulder pain, neck pain and/or osteoarthritis). Patients 18 years of age or older, who understand English, are experiencing chronic musculoskeletal pain for three months or more and have not received acupuncture therapy in the past 3 months will be invited to participate. We will recruit 120 outpatients with chronic pain from Mount Sinai Beth Israel's (MSBI) Family Medicine and other primary care practices. Referrals will be through primary care providers or by patient self-referral. The goal of this project is to develop a low-cost, effective integrative intervention for chronic pain which can be replicated in underserved settings across the U.S. The physician in charge of this study is Benjamin Kligler, M.D., M.P.H.

Eligible participants will be scheduled for a face-to-face interview, at which time consent will be obtained and baseline measures will be collected. Baseline measures include collecting demographic data and information on depression, pain/pain free days and medication use.

To follow, a 4-week run-in period where usual care is delivered will be held to establish baseline pain levels. During this time, participants will be contacted at 2-week intervals to complete a brief pain assessment. If a waiting list becomes necessary, delay may become longer.

Participants will then be invited to participate in an 8-week, group-based acupuncture treatment intervention delivered by a licensed acupuncturist. The group will meet weekly for 8 consecutive weeks, each session lasting about 75 minutes held at the Center for Health and Healing located at 245 Fifth Ave in Manhattan. Sessions will be held during evening and weekend hours to facilitate scheduling.

We will collect information on pain, pain symptoms, mood, function and analgesic use at 1, 8, 12 and 24 week(s) following the beginning of the intervention. We will collect this information in-person or by telephone as preferred by the participant. Participants will not receive an incentive to attend group sessions but will receive incentives at enrollment and for completing research interviews at 12 and 24 weeks following treatment intervention ($20 at each of these three time points).

While subject records are confidential, there may be loss of confidentiality due to the group acupuncture setting. Intervention risks are low: Acupuncture needles are pre-sterilized and inserted once only and then properly discarded. Acupuncture therapy is safe with a 'relative' risk that is low. The risks associated with providing protected health information (PHI) will be minimized by assigning a unique participant identification code (ID number) that will be used to identify all data reported for each participant. The study staff will store all PHI in a secure and protected site at the Center for Health and Healing. The study results will be stored in a locked cabinet and any study information stored in a computer will be password protected. Only the study staff will have access to the study results.

Subjects will be reminded of the elements of participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older, who understand English, are experiencing chronic musculoskeletal pain for three months or more and have not received acupuncture therapy in the past 3 months

Exclusion Criteria:

* Exclusion criteria will also include patients who have severe psychiatric problems as assessed by the study team (e.g., chronic interpersonal problems, cognitive impairment or active psychosis that is uncontrolled by medication that precludes the ability to provide informed consent or complete the survey instruments).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in pain symptoms | 24 weeks
  We will collect information on pain, pain symptoms, and analgesic use at 1, 8, 12 and 24 week(s) following the beginning of the intervention. We will collect this information in-person or by telephone as preferred by the participant.
Change in mood | up to 24 weeks
  We will collect information on mood at 1, 8, 12 and 24 week(s) following the beginning of the intervention. These measures will be collected by the use of validated tools which include scales and questionnaire such as BPI, CES-D and PGIC. We will track and see if our study interventions impact participants' mood
Change in analgesic use | up to 24 weeks
  We will collect information on pain, pain symptoms, and analgesic use at 1, 8, 12 and 24 week(s) following the beginning of the intervention. We will collect this information in-person or by telephone as preferred by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Kligler, MD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- The Center for Health and Healing, New York, New York, United States